CLINICAL TRIAL: NCT06469346
Title: Comparison Between Eccentric Exercise and Static Stretching on Hamstring Muscle Flexibility in Healthy Young
Brief Title: Comparison of Eccentric Exercise and Static Stretching on Muscle Flexibility
Acronym: COEESS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de La Frontera (Other)
Responsible Party: Principal Investigator, Gabriel Nasri Marzuca-Nassr, Professor, Universidad de La Frontera
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MGTFNG-2024
Record Dates: First submitted 2024-06-13; First posted 2024-06-21 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Muscle Stretching Exercise; Range of Motion, Articular
Keywords: Eccentric resistance exercise; Static Stretching; Muscle Flexibility; Range of Movement
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Eccentric Exercise Group (EEG) (Experimental): These participants will be subjected to 6 weeks of Nordic hamstring eccentric exercise (3 times per week)
  Interventions: Other: Nordic Hamstring Eccentric Exercise Training
- Static Stretching Group (SSG) (Experimental): These participants will be subjected to 6 weeks of passive static stretching on hamstring muscle (3 times per week)
  Interventions: Other: Passive Hamstring Static Stretching Training
- Control Group (Other): These participants will not be under any type of treatment during the intervention protocol
  Interventions: Other: Control Group

INTERVENTIONS:
Other: Nordic Hamstring Eccentric Exercise Training — Warm up: stationary bycicle at 50 watts and 60 bpm Mobility exercises for hip and knee joint
  Nordic eccentric exercise protocol:
  * Week 1: 2 sets x 5 repetitions
  * Week 2: 2 sets x 6 repetitions
  * Week 3: 3 sets x 6 repetitions
  * Week 4-6: 3 sets x 8 repetitions
  Arms: Eccentric Exercise Group (EEG)
Other: Passive Hamstring Static Stretching Training — Warm up: stationary bycicle at 50 watts and 60 bpm Mobility exercises for hip and knee joint
  * Week 1-2: 1 set x 2 repetitions of 30 seconds
  * Week 3: 1 set x 3 repetitions of 30 seconds
  * Week 4-6: 1 set x 3 reps of 40 seconds
  Arms: Static Stretching Group (SSG)
Other: Control Group — No intervention
  Arms: Control Group

SUMMARY:
Background: Muscle flexibility is a fundamental physical quality for body development, daily life and sports activities, and also for maintaining muscle quality during aging. Limited flexibility leads to an increased prevalence of musculoskeletal injury in general population and longer return to sports activities.

Among the existent strategies to increase muscle flexibility in sports training and physical rehabilitation, static stretching is commonly used by health and physical activity professionals. Its effectiveness in increasing flexibility has been widely demonstrated; however its effects on muscle strength and power remains controversial.

Therefore, eccentric resistance exercise has been proposed as an effective intervention for increasing muscle flexibility through structural changes on muscle architecture (pennation angle and fascicle length) with the additional benefit of resistance training on muscle strength and power. Nonetheless, its unknown if the increase in muscle flexibility through eccentric resistance exercise could be similar to what has been previously demonstrated with static stretching.

DETAILED DESCRIPTION:
Hypothesis: The increase in hamstring flexibility after 6 weeks of eccentric resistance training in young males would be similar compared to 6 weeks static stretching training in the same population.

Goals: The primary aim of the study is to compare the effectiveness of 6 weeks eccentric resistance training vs 6 weeks static stretching training on hamstring flexibility in young males.

Specific Goals: Determine the effect of 6 weeks excentric exercise training and 6 weeks static stretching training on unilateral maximal isometric voluntary strength between both groups

To compare the effect of 6 weeks excentric exercise training and 6 weeks static stretching training in structural changes on muscle architecture (pennation angle, fascicle length and muscle thickness).

Methodology:

Study design: Forty two young males between 18 and 35 years will be divided into three groups: hamstring eccentric resistance training group (EEG, n=14), hamstring static stretching group (SSG, n=14) and control group (CG, n=14). Volunteers of eccentric resistance training group will be subjected to 6 weeks of Nordic hamstring exercise (3x/wk), while volunteers of static stretching group will be subjected to 6 weeks of hamstring passive static stretching (3x/wk). Control group will not attend any type of intervention. Before and after 6 weeks of training, Knee Extension Angle and Sit and Reach test will be performed for measuring hamstring flexibility. Unilateral Hamstring Isometric Maximal Voluntary Strength will be determined by load cell force transducer, and pennation angle, fascicle length and muscle thickness of Long Head Biceps Femoris will be conducted through muscle ultrasonography

Study parameters/endpoint:

The main study endpoint is the increase in hamstring flexibility assessed with Knee Extension Angle and Sit and Reach Test.

Secondary endpoints include Unilateral Hamstring Isometric Maximal Voluntary Strength (IMVS) and Architectural changes in Long Head Biceps Femoris muscle.

Other parameters include age, body weight, body height, body mass index (BMI), level of physical activity.

Expected results: With the proposed project, the investigators expect that eccentric exercise training will increase hamstring muscle flexibility at similar level compared with static stretching training. The findings will define the potential of eccentric exercise training on muscle flexibility in healthy participants. These results could expand the benefits of this type of exercise training focused on being included in populations with limited mobility such as elderly and injured populations

ELIGIBILITY:
Inclusion Criteria:

* Masculine University students between 18 and 35 years old
* Physically Inactive considering physical activity recommendations from World Health Organization
* Bilateral hamstring muscle stiffness defined as <160° in passive Knee Extension Angle Test
* Body Max Index 18,5 < BMI < 24,9 kg/m2

Exclusion Criteria:

* Lower back and lower limb (hip, thigh, knee, ankle) musculoskeletal injury in the last 12 months.
* Hamstring injury (strain, tendinopathy, tendon avulsion) previously during the period of life
* Dietary anabolic supplements consumption
* Musculoskeletal, cardiovascular, respiratory o similar health condition that limits participation on physical activity programs
* Regular resistance training (2 or more times per week, carrying out progressive training) in the previous 6 months
* Smoker (1 cigarette per day)

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Estimated)
Dates: Start 2025-03-03 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Knee Extension Angle | Before and after 6 weeks of training
  The degree changes in passive knee extension will be assessed using Passive Knee Extension Angle Test after intervention
Sit-and-Reach | Before and after 6 weeks of training
  The distance (in centimeters) of change on functional posterior chain flexibility will be obtained in Sit-and-Reach Test after intervention

SECONDARY OUTCOMES:
Maximal Isometric Voluntary Strength | Before and after 6 weeks of training
  Change in unilateral isometric hamstring strength will be evaluated with load cell force transducer after intervention
Long Head Biceps Femoris Pennation Angle | Before and after 6 weeks of training
  Change in pennation angle will be measured using muscular ultrasound after intervention
Long Head Biceps Femoris Fascicle Length | Before and after 6 weeks of training
  Change in fascicle length will be measured using muscular ultrasound after intervention
Long Head Biceps Femoris Muscle Thickness | Before and after 6 weeks of training
  Change in muscle thickness will be measured using muscular ultrasound after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel N Marzuca-Nassr, Principal Investigator — Universidad de La Frontera
Locations (1):
- Universidad de La Frontera, Temuco, Cautín, Chile

IPD SHARING:
Plan to Share IPD: Undecided